CLINICAL TRIAL: NCT03362242
Title: A Phase 1 Single and Multiple Dose-Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Effect of ARO-AAT on Serum Alpha-1 Antitrypsin Levels in Normal Adult Volunteers
Brief Title: Study of ARO-AAT in Normal Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AROAAT1001
Record Dates: First submitted 2017-11-30; First posted 2017-12-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARO-AAT (Active Comparator)
  Interventions: Drug: ARO-AAT Injection
- Placebo (Placebo Comparator)
  Interventions: Other: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: ARO-AAT Injection — Single or multiple doses of ARO-AAT by subcutaneous (sc) injections
  Arms: ARO-AAT
Other: Sterile Normal Saline (0.9% NaCl) — Calculated volume to match active comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single- and multiple-ascending doses of ARO-AAT in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Women of child bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be willing to use contraception
* Willing to provide written informed consent and to comply with study requirements
* Non-smoker for at least one year
* Normal lung function
* No abnormal finding of clinical relevance at Screening
* Normal AAT level at Screening visit

Exclusion Criteria:

* Clinically significant health concerns
* Regular use of alcohol within one month prior to Screening
* Use of an investigational agent or device within 30 days prior to dosing or current participation in an investigational study
* Recent use of illicit drugs
* Use of any drugs or dietary/herbal supplements know to interfere with liver metabolism

NOTE: additional inclusion/exclusion criteria may apply, per protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) Possibly or Probably Related to Treatment | Part A (single-ascending dose [SAD] phase): up to 29 (+/- 2) days post-dose; Part B (multiple-ascending dose [MAD] phase): up to 113 (+/- 2) days post-dose

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ARO-AAT: Maximum Observed Plasma Concentration (Cmax) | Part A (single-ascending dose [SAD] phase): up to 48 hours post-dose; Part B (multiple-ascending dose [MAD] phase): up to 48 hours post-dose
PK of ARO-AAT: Time to Maximum Plasma Concentration (Tmax) | Part A (SAD phase): up to 48 hours post-dose; Part B (MAD phase): up to 48 hours post-dose
PK of ARO-AAT: Terminal Elimination Half-Life (t½) | Part A (SAD phase): up to 48 hours post-dose; Part B (MAD phase): up to 48 hours post-dose
PK of ARO-AAT: Area Under the Plasma Concentration Versus Time Curve From Zero to 24 Hours (AUC0-24) | Part A (SAD phase): up to 48 hours post-dose; Part B (MAD phase): up to 48 hours post-dose
PK of ARO-AAT: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUCinf) | Part A (SAD phase): up to 48 hours post-dose; Part B (MAD phase): up to 48 hours post-dose
Percent Change in Serum Alpha-1 Antitrypsin (AAT) Levels From Day 1 Pre-Dose Baseline to Nadir | Part A (SAD phase): up to 29 (+/- 2) days; Part B (MAD phase): up to 113 (+/- 2) days
Duration of Response of Serum AAT levels From Nadir Back to Above 20% of Baseline or Above 90 mg/dL | Part A (SAD phase): up to 29 (+/- 2) days; Part B (MAD phase): up to 113 (+/- 2) days

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site 1, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No